CLINICAL TRIAL: NCT05701137
Title: Effectiveness of an Eye Movement Desensitization and Reprocessing (EMDR) Intervention for the Prevention of Post-traumatic Symptoms in Perinatal Loss
Brief Title: Effectiveness of an EMDR Intervention for Perinatal Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: EMDR Europe (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022-03
Record Dates: First submitted 2022-12-19; First posted 2023-01-27 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-03

CONDITIONS: Pregnancy Loss; PTSD
Keywords: perinatal loss; PTSD; EMDR
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EMDR-RTE (Experimental): Eye movement desensitization and reprocessing in its recent traumatic episode version.
  Interventions: Other: EMDR-RTE
- TAU (Active Comparator): Usual treatment by a psychologist.
  Interventions: Other: TAU

INTERVENTIONS:
Other: EMDR-RTE — The experimental group will have EMDR recent traumatic event.
  Arms: EMDR-RTE
Other: TAU — The comparator group will have usual psychological intervention.
  Arms: TAU

SUMMARY:
The investigators objectives is to assess the effectiveness of Eye Movement Desensitization and Reprocessing - recent traumatic episode (EMDR-RTE) as a preventive intervention for Posttraumatic Stress Disorder (PTSD) symptoms after perinatal loss.

The hypothesis is that EMDR-RTE treatment may prevent post-traumatic and depressive symptoms in women who suffered perinatal loss.

DETAILED DESCRIPTION:
Perinatal loss is a general term that refers to a loss from conception to one month postpartum. It is a grief that is still socially unauthorized, however, it is a situation with significant traumatic potential. However, there are no studies evaluating the effectiveness of Eye Movement Desensitization and Reprocessing (EMDR) for the prevention or treatment of perinatal loss. We propose an one-site, open label, randomized controlled trial with the aim of assessing the effectiveness of EMDR recent traumatic episode (EMDR-RTE) as a preventive intervention for PTSD symptoms after perinatal loss. A total of 40 women who have suffered a perinatal loss from the Maternal-Fetal Medicine Service of a tertiary university hospital will be recruited. Women will be randomized to EMDR-RTE or treatment as usual (TAU). Researchers will compare EMDR-RTE and TAU to see if women receiving EMDR-RTE treatment had lower levels of post-traumatic and depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* be over 18 years old
* agree to participate and sign the informed consent
* request psychological treatment

Exclusion Criteria:

* active substance use disorder
* cognitive disability
* language barrier

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-03-23 (Actual)

PRIMARY OUTCOMES:
PCL-5 | Within the first month after perinatal loss
  PTSD Checklist for DSM-5
PCL-5 | 3 months after perinatal loss
  PTSD Checklist for DSM-5

SECONDARY OUTCOMES:
STAI S/T | Within the first month after perinatal loss
  Spielberger State/Trait Anxiety Inventory
STAI S/T | 3 months after perinatal loss
  Spielberger State/Trait Anxiety Inventory
BDI-II | Within the first month after perinatal loss
  Beck Depression Inventory
BDI-II | 3 months after perinatal loss
  Beck Depression Inventory

OTHER OUTCOMES:
Satisfaction survey | 3 months after perinatal loss

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic sede Maternitat, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Sureda-Caldentey B, Garcia-Gibert C, Martinez A, Gimenez Y, Segu X, Mallorqui A, Gelabert E, Roca-Lecumberri A, Torres-Gimenez A. Effectiveness of an eye movement desensitization and reprocessing intervention for the prevention of post- traumatic symptoms in perinatal loss: a randomized pilot controlled trial. Front Psychiatry. 2025 Jun 9;16:1593306. doi: 10.3389/fpsyt.2025.1593306. eCollection 2025. PMID 40551815